CLINICAL TRIAL: NCT04125264
Title: The Application of Intense Therapeutic Ultrasound in Plantar Fasciitis. A Randomized, Non-probabilistic and Superiority Controlled Clinical Trial
Brief Title: Intense Therapeutic Ultrasound (ITU) to Treat Plantar Fasciitis
Acronym: ITU
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Universidad Complutense de Madrid (Other)
Responsible Party: Principal Investigator, Raúl Juan Molines Barroso, Phd, Clinical Professor, Universidad Complutense de Madrid
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 18/399-R_P
Record Dates: First submitted 2019-10-10; First posted 2019-10-14 (Actual); Last update posted 2019-10-16 (Actual); Status verified 2019-10

CONDITIONS: Plantar Fasciitis; Plantar Fasciitis, Chronic; Ultrasound Therapy
MeSH Terms: conditions — Fasciitis, Plantar

STUDY DESIGN:
Intervention Model Description: Randomized, Non-probabilistic and Superiority Controlled Clinical Trial.
Masking Description: Patient located in experimental group will be treated with ITU. Patient located in control group will be treated with the same protocoll of ITU without intensity.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Intense therapeutic Ultrasound (Experimental): During the trial two applications of 1000 pulses each one (day one and day thirty) will be applied. Pulse regulation could be modified from 4 to 5 joules depending the presence or not of pain.
  Conservative treatment of plantar fasciitis include: custom made foot orthosis with the same general characteristics plus plantar fasciia and achilles tendon stretching.
  Interventions: Device: Intense Therapeutic Ultrasound
- Control group (No Intervention): Non ITU application. Conservative treatment of plantar fasciitis include: custom made foot orthosis with the same general characteristics plus plantar fasciia and achilles tendon stretching.

INTERVENTIONS:
Device: Intense Therapeutic Ultrasound — Application of 1000 pulses, until 5000 joules (5 joules per pulse), during approximately 15 minutes, with the possibility of 5 minutes rest, depending on the tolerance of the patient.
  Arms: Intense therapeutic Ultrasound

SUMMARY:
It was previously hypothesized that patients receiving Intense Therapeutic Ultrasound (ITU) in addition to the standard of care would have a more rapid resolution of pain, faster return to activities, and a decrease in intra- and perifascial lesions.

DETAILED DESCRIPTION:
Intense Therapeutic Ultrasound (ITU) is an established ultrasound-based therapy in which sound waves are concentrated and focused into a well-defined specific area of musculoskeletal tissue. Previous researches hipothesize that the application of ITU improve and accelerate healing in patients with chronic plantar fasciitis.

ELIGIBILITY:
Inclusion Criteria:

* Both sex patients.
* Plantar fasciitis diagnosis: pain during walking during the first steps in the morning; pain due to palpation of plantar fasciia insertion.
* Chronic pain of at least 6 month.
* Longitudinal thickness of the plantar fasciia more than 4 millimeters.
* No previous surgery in the plantar fasciia.
* No previous application of alternative treatments such us shock waves or injections (last ninety days)

Exclusion Criteria:

* Platelet count disorder or anticoagulation therapy.
* Anti-inflammatories usual treatment for the treatment of plantar fasciitis.
* Diabetic foot syndrome.
* Presence of metabolic disease such us: hypertension, hiper or hipothyroidism.
* Pregnancy or breastfeeding.
* Previous treatment with fluoroquinolones antibiotic.
* Bilateral plantar fasciitis.
* Diagnosed Autoimmune disesase.
* Morphofunctional disorders in the foot and ankle.
* Diagnosed fibromyalgia.
* Heel disestesy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2019-10 (Estimated); Primary Completion 2020-10 (Estimated); Study Completion 2021-10 (Estimated)

PRIMARY OUTCOMES:
Pain reduction | 24 weeks
  Use of a Subjective Visual Analogue Scale (SVAS): the outmost left (0 cm) was labelled pain absence and the outmost right (10 cm) was labelled the maximum imagined pain.
Plantar fasciia thickness reduction | 24 weeks
  Longitudinal view of the plantar fasciia with the use of ultrasound probe.

SECONDARY OUTCOMES:
Hypoechoic volume area reduction | 24 weeks
  Longitudinal and transversal view of the hypoechoic area of plantar fasciia with the use of ultrasound probe.
Ankle range of motion reduction | 24 weeks
  Goniometry of the ankle in the extended and flexed position of the knee
Time to incorporation to daily live activities | 24 weeks
  Patients satisfaction scale (6 items)
Autonomous gait without pain in the heel | 24 weeks
  Patients autonomous gait scale (6 items)
Improvement of patients satisfaction | 24 weeks
  Patients satisfaction scale (6 items)

CONTACTS AND LOCATIONS:
Overall Officials: José Luis Lázaro Martínez, Phd, Principal Investigator — Universidad Complutense Madrid
Locations (1):
- Diabetic foot Unit Complutense University, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No